CLINICAL TRIAL: NCT01629069
Title: A Resilience Intervention Involving Mindfulness Training for Transplant and Cancer Patients and Their Caregivers
Brief Title: A Transplant or Cancer Resilience Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cynthia M. Stonnington, M.D., Chair, Department of Psychiatry & Psychology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-004988
Record Dates: First submitted 2012-06-21; First posted 2012-06-27 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Behavior; Emotions
Keywords: stress; mindfulness; coping
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participant in MBRT (Active Comparator): 6 sessions of Mindfulness Based Resilience Training
  Interventions: Behavioral: Mindfulness based Resilience Training

INTERVENTIONS:
Behavioral: Mindfulness based Resilience Training — 6 weekly group sessions

SUMMARY:
The overall aim of this protocol is to examine patient and care-giver outcomes and acceptance of a new 6 week intervention in Arizona for our transplant and cancer patients and their care-givers, designed to improve quality of life, decrease perceived stress, and improve medical outcomes, that has been approved as a pilot clinical program at Mayo Clinic in Arizona.

DETAILED DESCRIPTION:
Transplant medicine and cancer are major strategic foci of Mayo Clinic. At Mayo Clinic, we are often challenged to respond adequately to the high levels of stress encountered by our transplant patients and their care-givers. The overall aim of this project is to pilot a 6 session intervention in Arizona for our transplant and cancer patients and their care-givers, designed to improve quality of life, decrease perceived stress, and improve medical outcomes. Demonstration of a feasible and effective program will allow us to offer similar programs at all three sites. This program has potential to better meet our transplant patients' needs, improve outcomes, and set us apart from other transplant programs who do not offer this intervention for patients and caregivers. Psychiatry already has a good collaboration with transplant medicine, with psychiatry screening transplant patients and following a large subset of patients. Many of the referrals to psychiatry post-transplant have to do with difficulty managing stress or break-down in care-giver support. The proposed program would address this unmet need with a more comprehensive intervention than is currently available at the Mayo Clinic. The role of this pilot program is to:

* Explore the feasibility of routinely offering a resilience intervention involving mindfulness based stress reduction to our solid organ and stem-cell transplant and cancer patients and their care-givers.
* Pilot a mindfulness-based group treatment for stress reduction to assess its impact, using standardized rating tools, on transplant patient stress-levels, sleep quality, anxiety, depression, medical outcomes, and health-care utilization
* Examine patient and care-giver acceptance/adherence and satisfaction
* Understand the resources both in terms of staffing and fees required to offer this as a clinical program in the future
* Explore the reimbursement options for covering the program's expenses.

ELIGIBILITY:
Inclusion Criteria:

* Patient listed for liver, heart, kidney, or bone marrow transplant
* Patient who has received a liver, heart, kidney, or bone marrow transplant
* Caregiver of transplant patient
* patient with diagnosis of cancer, either active or in remission
* supportive care partner of cancer patient

Exclusion Criteria

* Suicidal
* Severe cognitive impairment
* psychotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Patient questionaire | baseline to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Stonnington, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States